CLINICAL TRIAL: NCT06032052
Title: Prospective, Single-arm Phase II Clinical Study of Single-drug Chemotherapy Plus Immunotherapy in Metastatic Non-small Cell Lung Cancer Elderly Patients
Brief Title: Single-drug Chemotherapy Plus Immunotherapy in Metastatic Non-small Cell Lung Cancer Elderly Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Chief physician, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Unicorn
Record Dates: First submitted 2023-08-22; First posted 2023-09-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Elderly Patients; Metastatic Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic NSCLC patients over 65 years old (Experimental): In metastatic NSCLC patients over 65 years old, we employed gemcitabine or paclitaxel or vinorelbine plus immunotherapy for squamous cell carcinoma. Paclitaxel or pemetrexed plus immunotherapy are available for non-squamous and non-small cell lung cancer.
  Interventions: Drug: Single drug chemotherapy plus immunotherapy

INTERVENTIONS:
Drug: Single drug chemotherapy plus immunotherapy — The choice of chemotherapy plus immunotherapy for squamous cell carcinoma is gemcitabine or paclitaxel or vinorelbine. Paclitaxel or pemetrexed are available for monotherapy for non-squamous and non-small cell lung cancer. Immunotherapy drugs can be Pembrolizumab /Penpulimab/ Camrelizumab/ Tislelizumab / Sintilimab/ sulgarizumab and so on
  Other Names: monochemotherapy plus immunotherapy

SUMMARY:
Lung cancer is the cancer with the highest morbidity and mortality among men in the world. The proportion of elderly lung cancer patients in the global lung cancer population is steadily increasing, at the same time, it is also the age group with the highest lung cancer mortality, but there is little evidence for treatment of elderly lung cancer patients. In this study, the investigators set the definition of the elderly to 65 years and older.

The progression-free survival (PFS) and overall survival (OS) of immunotherapy plus chemotherapy were higher than those of chemotherapy alone, which established the dominant position of dual-drug chemotherapy combined with immunotherapy. Studies showed that elderly patients benefit from immunotherapy.

It is controversial whether elderly advanced non-small-cell-lung-cancer (NSCLC) patients should receive single-drug chemotherapy or dual-drug chemotherapy. MILES-3 and MILES-4 studies show that in the advanced NSCLC elderly patients, combined with cisplatin on the basis of single drug chemotherapy can not significantly prolong OS, and can not improve the overall health status of patients. Based on the results of this study, single drug chemotherapy is still the preferred first-line regimen. Another study showed that carboplatin combined with paclitaxel had longer OS than gemcitabine or vinorelbine alone in elderly patients with advanced NSCLC with a performance status (PS) score of less than 2. In the era of immunotherapy, it is not clear whether single-drug chemotherapy combined with immunotherapy can achieve the same therapeutic effect as dual-drug chemotherapy combined with immunotherapy. Therefore, the purpose of this study is to investigate the efficacy and safety of single-drug chemotherapy plus immunotherapy in elderly metastatic NSCLC patients.

DETAILED DESCRIPTION:
Lung cancer is the cancer with the highest morbidity and mortality among men in the world. The age range in which lung cancer is most commonly diagnosed is 65-74 years old. The proportion of elderly lung cancer patients in the global lung cancer population is steadily increasing, at the same time, it is also the age group with the highest lung cancer mortality, but there is little evidence for treatment of elderly lung cancer patients. The investigators pay special attention to elderly patients because they are a unique group.

With regard to the definition of "elderly", considering that more than half of cancer patients are aged 65 or above. Therefore, we set the definition of the elderly in this phase II clinical study to 65 years and older.

The results of Keynote-042 study, Keynote-189 study and Keynote-407 study all showed that the progression-free survival (PFS) and overall survival (OS) of immunotherapy plus chemotherapy were higher than those of chemotherapy alone, which established the dominant position of dual-drug chemotherapy combined with immunotherapy. Meta analysis showed that in patients with advanced NSCLC, immunotherapy prolonged OS and PFS compared with chemotherapy, and the prolongation of PFS was not related to age, while OS also benefited in patients aged 65 to 75 years. To sum up, elderly patients benefit from immunotherapy.

It is controversial whether elderly advanced NSCLC patients should receive single-drug chemotherapy or dual-drug chemotherapy. MILES-3 and MILES-4 studies show that in the advanced NSCLC elderly patients, combined with cisplatin on the basis of single drug chemotherapy can not significantly prolong OS, and can not improve the overall health status of patients. Based on the results of this study, single drug chemotherapy is still the preferred first-line regimen. Another study showed that carboplatin combined with paclitaxel had longer OS than gemcitabine or vinorelbine alone in elderly patients with advanced NSCLC with a PS score of less than 2. In the era of immunotherapy, it is not clear whether single-drug chemotherapy combined with immunotherapy can achieve the same therapeutic effect as dual-drug chemotherapy combined with immunotherapy. Therefore, the purpose of this study is to investigate the efficacy and safety of single-drug chemotherapy plus immunotherapy in elderly metastatic NSCLC patients, in order to reduce the adverse reactions without reducing the curative effect and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Regardless of sex, age ≥ 65, PS 0-2.
2. metastatic NSCLC of American Joint Committee on Cancer (AJCC) 8th edition confirmed by histology or cytology.
3. No mutation or fusion of common driving genes, such as epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), ROS proto-oncogene 1 (ROS-1).

   (adenocarcinoma requires genetic testing).
4. Positive expression of Programmed cell death 1 ligand 1（PD-L1） (TPS ≥ 1%).
5. First-line treatment (stable brain or bone metastasis, or stable symptoms after local treatment).
6. Before treatment, there were perfect enhanced CT images of chest and supraclavicular area, and measurable tumor lesions.
7. The estimated survival time is not less than 6 months.
8. The clinical laboratory criteria within 2 weeks before treatment are as follows: hemoglobin ≥ 110g / L, leukocytes ≥ 4x109 / L, platelet ≥ 100x109 / L, liver and kidney function indexes (such as glutamic pyruvic transaminase, glutamic oxaloacetic transaminase, urea nitrogen, creatinine) were all within 1.25 times of the upper limit of the normal value.
9. Informed understanding and voluntary participation in this study, and informed consent has been signed.

Exclusion Criteria:

1. Mutation or fusion of common driving genes (EGFR,ALK or ROS1).
2. Have received systemic treatment before.
3. Previous suffering from other malignant tumors (except stage I non-melanotic skin cancer or cervical carcinoma in situ) or other malignant tumors at the same time.
4. Other drugs are being tested.
5. Patients with positive HIV and are receiving antiviral therapy .
6. Active pulmonary tuberculosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | up to 12 months
Objective response rate | up to 6 months

SECONDARY OUTCOMES:
Overall survival | up to 18 months
Disease control rate | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Han, Principal Investigator — Hubei Cancer Hospital
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes